CLINICAL TRIAL: NCT04227756
Title: Comparative Acute Effects of LSD, Psilocybin and Mescaline in a Random-Order Placebo-Controlled Cross-Over Study in Healthy Subjects
Brief Title: Comparative Acute Effects of LSD, Psilocybin and Mescaline
Acronym: LPM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BASEC 2019-02023
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide; Psilocybin; Mescaline

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, 4-period cross-over design with four treatment conditions
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LSD-100 (Experimental): Cross-over within-subject design with all treatment conditions, separated by a wash-out phase of at least 10 days
  Interventions: Drug: LSD
- Psilocybin-20 (Active Comparator): Cross-over within-subject design with all treatment conditions, separated by a wash-out phase of at least 10 days
  Interventions: Drug: Psilocybin
- Mescaline-300/500 (Active Comparator): Cross-over within-subject design with all treatment conditions, separated by a wash-out phase of at least 10 days
  Interventions: Drug: Mescaline
- Placebo (Placebo Comparator): Cross-over within-subject design with all treatment conditions, separated by a wash-out phase of at least 10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LSD — LSD 0.1 mg per os, single dose OR Psilocybin 20 mg per os, single dose OR Mescaline 300 mg per os, single dose OR Placebo
  Arms: LSD-100
Drug: Psilocybin — Psilocybin 20 mg per os, single dose
  Arms: Psilocybin-20
Drug: Mescaline — Mescaline 300 mg or 500 mg per os, single dose
  Arms: Mescaline-300/500
Other: Placebo — Placebo (Mannitol)
  Arms: Placebo

SUMMARY:
LSD, psilocybin and mescaline are widely used for recreational and ethnomedical purposes. All three substances are thought to induce prototypical psychedelic effects primarily via stimulation of the 5-HT2A receptor. However, there are differences in the substances' molecular structures and receptor activation profiles which may induce differential subjective effects. To date, there are no modern studies comparing LSD, psilocybin and mescaline directly within the same clinical study and research subjects using validated psychometric tools. Therefore, the LPM-Study compares the acute effects of LSD, psilocybin, mescaline and placebo in a double-blind, placebo-controlled, 4-period cross-over design with four treatment conditions: 1) 100 μg LSD, 2) 20 mg psilocybin, 3) 300 or 500 mg mescaline, and 4) placebo.

DETAILED DESCRIPTION:
LSD (lysergic acid diethylamide), psilocybin (the active substance in "magic mushrooms") and mescaline (the active substance in Peyote and San Pedro cacti) are serotonergic hallucinogens widely used for recreational and/or ethnomedical purposes. LSD, psilocybin and mescaline are thought to induce prototypical psychedelic effects primarily via stimulation of the 5-HT2A receptor. However, there are differences in their molecular structures (LSD: ergoline, psilocybin: tryptamine; mescaline: phenethylamine)and receptor activation profiles which may induce different subjective effects. To date, there are no modern studies comparing these three substances directly within the same clinical study and research subjects using validated psychometric tools. Therefore, the LPM-Study compares the acute effects of LSD, psilocybin, mescaline and placebo in a double-blind, placebo-controlled, 4-period cross-over design with four treatment conditions: 1) 100 μg LSD, 2) 20 mg psilocybin, 3) 300 or 500 mg mescaline, and 4) placebo. The main objective of this study is to determine whether LSD, psilocybin and mescaline produce qualitatively similar subjective alterations of mind and associated brain activity patterns despite their unique receptor activation profiles. The study investigates psychological (psychometry), physiological and neuronal (magnetic resonance imaging) variables. The LPM-Study provides insight into the acute effects profiles of three serotonergic hallucinogens. It will enhance the understanding of psychedelic-induced altered states of consciousness in humans and will be relevant for the fields of psychiatry, psychology, and forensic toxicology.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids from the evenings prior to the study sessions to the end of the study days
7. Willing not to operate heavy machinery within 48 hours after substance administration
8. Willing to use double-barrier birth control throughout study participation
9. Body mass index between 18-29 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Hallucinogenic substance use (not including cannabis) more than 20 times or any time within the previous two months
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)
11. Failure of MRI-related criteria

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
5 Dimensions of Altered States of Consciousness (5D-ASC) | 18 months
  5D-ASC subscale ratios
fMRI resting state functional connectivity (RSFC) | 18 months
  Spontaneous low-frequency fluctuations in BOLD signal during resting state

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 18 months
  Assesses the intensity and duration of subjective effects on a scale from 0% - 100% with higher scores representing more intense effects
States of Consciousness questionnaire (SCQ) | 18 months
  Assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely")
Blood pressure | 18 months
  Assessment of sympathetic activation
Heart rate | 18 months
  Assessment of sympathetic activation
Body temperature | 18 months
  Assessment of sympathetic activation
Pupil size | 18 months
  Assessment of sympathetic activation
Drug plasma levels | 18 months
  Plasma levels of investigational drugs
Oxytocin levels | 18 months
  Levels of oxytocin in blood plasma
Blood-derived neurotrophic factor (BDNF) | 18 months
  Blood plasma levels of BDNF
Renal clearance values | 18 months
  Renal clearance values of investigational drugs through urine recovery
NEO-Five-Factor-Inventory (NEO-FFI) | 18 months
  Assesses personality traits
Freiburger Persönlichkeitsinventar (FPI) | 18 months
  Assesses personality traits
Saarbrücker Persönlichkeitsfragebogen (SPF) | 18 months
  Assesses personality traits
Adjective Mood Rating Scale (AMRS) | 18 months
  Assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely"
Mysticism Scale (MS) | 18 months
  Assesses the occurrence and intensity of mystical qualities in altered states of consciousness on a 9-point Likert scale ranging from -4 ("extremely inapplicable") to +4 ("extremely applicable"), with higher values indicating a more intense experience
Elliot Humility Scale (EHS) | 18 months
  Assesses the personality trait humility through 13 items on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree"
Jankowski Humility Scale (JHS) | 18 months
  Assesses the personality trait humility through 18 items on a 5-point Likert scale ranging from "not at all" to "strongly"
Arnett Inventory of Sensation Seeking (AISS-d) | 18 months
  Assesses personality traits

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E. Liechti, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinical Trial Unit, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller L, Klaiber A, Ley L, Becker AM, Thomann J, Luethi D, Schmid Y, Liechti ME. Pharmacokinetics, Pharmacodynamics, and Urinary Recovery of Oral Mescaline Hydrochloride in Healthy Participants. Clin Pharmacokinet. 2025 Oct;64(10):1495-1506. doi: 10.1007/s40262-025-01544-x. Epub 2025 Jul 14. PMID 40658345
- [Derived] Ley L, Holze F, Arikci D, Becker AM, Straumann I, Klaiber A, Coviello F, Dierbach S, Thomann J, Duthaler U, Luethi D, Varghese N, Eckert A, Liechti ME. Comparative acute effects of mescaline, lysergic acid diethylamide, and psilocybin in a randomized, double-blind, placebo-controlled cross-over study in healthy participants. Neuropsychopharmacology. 2023 Oct;48(11):1659-1667. doi: 10.1038/s41386-023-01607-2. Epub 2023 May 25. PMID 37231080